CLINICAL TRIAL: NCT05091710
Title: Pilot Trial of a Community Health Worker Intervention to Improve Heart Failure Care in Rural Haiti
Brief Title: Haiti Community Health Workers (CHW) Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-41758; 1K23HL140133-01A1 (NIH)
Record Dates: First submitted 2021-09-15; First posted 2021-10-25 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Community health worker (CHW); ADAPT-ITT; Haiti
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Follow up care program for HF patients (Experimental): Discharged HF patients in rural Haiti will be receive a follow-up care program delivered by trained community health workers (CHWs).
  Interventions: Other: HF follow up care
- Standard of care (Other): Historical reference group who received standard of care for HF identified prior to CHW training.
  Interventions: Other: HF Standard of Care (SOC)

INTERVENTIONS:
Other: HF follow up care — The intervention will consist of follow up phone calls and visits during which the CHWs will remind patients about upcoming visits, ensure patient has sufficient medications, review medication schedule and provide education as needed.
  Arms: Follow up care program for HF patients
Other: HF Standard of Care (SOC) — SOC after discharge for HF is to notify patients of a follow-up visit at the hospital/clinic - about 7 days after discharge and provide patients about 30 days of medications at discharge. If a patient does not return for a follow-up appointment, there are no systems to track this missed visit, or to trigger active attempts to contact patients. For patients who come back to their scheduled 7-day visit, there is generally a 14-day visit followed by a 28-day visit.
  Arms: Standard of care

SUMMARY:
Evidence-based interventions to improve linkage and outcomes for heart failure (HF) patients requires input from stakeholders: patients, community health workers (CHWs), healthcare staff, and health system administrators.

In this research the investigators will assess a CHW intervention designed to improve linkage to care for HF patients. This intervention was systematically adapted for use in rural Haiti in a prior study using the Assessment, Decisions, Administration, Production, Topical Experts, Integration, Training staff, Testing (ADAPT-ITT) framework. The ADAPT-ITT framework provides 8 sequential phases to adapt interventions and programs to new target audiences. It has been applied successfully to the adaptation of several interventions for HIV among under-resourced communities leading to randomized clinical trials. With the first 6 steps of the ADAPT-ITT framework completed in a prior study, this protocol outlines the training and testing of the adapted CHW intervention.

In addition to assessing the feasibility, appropriateness, and acceptability of the adapted intervention through participants' feedback, the investigators will assess its efficacy in improving HF outcomes. The proposed intervention is targeted at both the patient domain - through improved peer support - and health system domain - by improving health system navigation.

DETAILED DESCRIPTION:
This is a clinical trial involving the training of 6 CHWs in a linkage-to-care intervention and the testing of the intervention on 30 HF patients. In a prior study, the ADAPT-ITT framework was used to adapt a CHW-based intervention for post-discharge HF patients in Haiti. This study represents the last two phases of the ADAPT-ITT framework: Training and Testing.

The study population will include adult HF patients (> 18 years of age), hospitalized for more than 48 hours, discharged from Hôpital-Universitaire de Mirebalais (HUM), without a prior clinic visit, living in Mirebalais Commune. Patients will be recruited for study participation shortly before discharge. A comparison group of 30 HF patients will be recruited and will not participate in the follow up care intervention. Those patients will be retrospectively identified from the medical record. The comparison group and will not receive any intervention. Six experienced CHWs will be trained to conduct the linkage to care intervention.

The intervention will include study visits in the form of home visits and phone calls performed by CHWs during which they will remind patients about upcoming visits, ensure patient has sufficient medications, review medication schedule and provide education as needed.

ELIGIBILITY:
Inclusion Criteria for patient participant:

* Adult HF patients
* Hospitalized >48 hours at Hôpital-Universitaire de Mirebalais (HUM)
* Anticipated discharge from HUM within 1-3 days
* Living in Mirebalais Commune, Haiti Inclusion criteria for historical patient reference group
* Adult HF patients
* Hospitalized >48 hours at HUM
* Discharged from HUM within the 12 months preceding the intervention
* Living in Mirebalais Commune

Exclusion Criteria for patient participant and historical patient reference group:

* None

Inclusion Criteria for CHW

* Adult
* Provide inpatient or outpatient care to HF patients
* Working in in Mirebalais

Exclusion Criteria for CHW

* None

Inclusion criteria for healthcare staff (provider/administrator)

* Hospital leadership involved in supervision of clinical care programs (i.e. Chief Executive Officer, Chief Medical Officer, Chief Operations Officer, Chief Nursing Officer, etc.)
* Leaders of the Community Health Department - including the nurse Director of Community Health, and Community Health Worker Supervisors.
* Healthcare providers at HUM involved in the care of patients with heart failure (i.e. internal medicine physicians, inpatient hospital nurses, outpatient clinic physicians, outpatient clinic nurses, etc.)

Exclusion criteria for healthcare staff (provider/administrator)

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of HF follow up program to patients | 90 days
  Acceptability of the HF follow up program to patients will be assessed using a 5-point Likert scale response to the question "Was it acceptable to have a CHW come to your home to educate you in your heart failure care and encourage clinic follow-up?" where 1=not acceptable, 5=very acceptable.
Acceptability of HF follow up program to Community Health Workers (CHWs) | 12 months
  Acceptability of the HF follow up program to CHWs will be assessed using a 5-point Likert scale response to the question "Was it acceptable to have a CHW come to your home to educate you in your heart failure care and encourage clinic follow-up?" where 1=not acceptable, 5=very acceptable.
Acceptability of HF follow up program to nurses/doctors | 12 months
  Acceptability of the HF follow up program to nurses/doctors will be assessed using a 5-point Likert scale response to the question "Was it acceptable to have a CHW come to your home to educate you in your heart failure care and encourage clinic follow-up?" where 1=not acceptable, 5=very acceptable.
Appropriateness of HF follow up program to patients | 90 days
  Appropriateness of HF follow up program to patients will be assessed using a 5-point Likert scale response to the question "Were you satisfied with the CHWs interactions with you?" where 1=not acceptable, 5=very acceptable.
Appropriateness of HF follow up program to CHWs | 12 months
  Appropriateness of HF follow up program to CHWs will be assessed using a 5-point Likert scale response to the question "Were you satisfied with the CHWs interactions with you?" where 1=not acceptable, 5=very acceptable.
Appropriateness of HF follow up program to nurses/doctors | 12 months
  Appropriateness of HF follow up program to nurses/doctors will be assessed using a 5-point Likert scale response to the question "Were you satisfied with the CHWs interactions with you?" where 1=not acceptable, 5=very acceptable.
Feasibility of HF follow up program to patients | 90 days
  Feasibility of HF follow up program to patients will be assessed by the percent of invited eligible patients who consent to participate. The higher the percentage of consenting patients, the more feasible the program.
Feasibility of HF follow up program to CHWs | 90 days
  Feasibility of HF follow up program to CHWs will be assessed by the percent of invited CHWs who complete the training. The higher the percentage, the more feasible the program.
Fidelity of HF follow up program | 90 days
  Fidelity of HF follow up program will be assessed by the percent of home visit checklist items completed by CHWs. The higher the percentage, the greater the fidelity.
HF follow up program intervention components delivered | 90 days
  Assessed by the number of interventions delivered based abstracted from the home visit checklist completed by the CHWs.
Completion of scheduled visits | 90 days
  Assessed by the percent of scheduled visits that were completed from the CHW records.
Percent of visits with all home visit checklist items completed | 90 days
  Assessed by dividing the number of visits with all home visit checklist items completed by the total number of visits.

SECONDARY OUTCOMES:
Linkage of HF patients | 30 days
  Percent of patients that complete 30 day follow up visit
Retention of HF patients | 90 days
  Percent of patients that complete 90 day follow up visit
Hospital readmission rate | 90 days
  Percent of patients that are readmitted to the hospital abstracted from the medical charts
Patient symptoms based on the New York Heart Association (NYHA) Classification | 90 days
  A New York Heart Association (NHYA) class from 1 to 4 will be assigned to each patient. The higher the classification the more serious the symptoms
  NYHA Classification - The Stages of Heart Failure:
  Class 1 - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class 2 - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class 3 - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class 4 - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Patient quality of life assessed European Quality of Life 5D (EuroQol 5D) | 30 days, 90 days
  Quality of life of patients will be assessed with the European Quality of Life 5D (EuroQol 5D) level. ThevEuropean Quality (EQ)-5D descriptive system is a preference-based Health-related quality of life (HRQL) measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to EQ-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Symptoms and quality of life based on the Kansas City Cardiomyopathy Questionnaire (KCCQ) | 30 days, 90 days
  The KCCQ will be used to assess symptoms, physical and social limitations, and quality of life in HF patients. Scores are scaled from 0 to 100 and will be summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.
Mortality rate in HF patients | 90 days
  The number of HF patients who die within 90 days following discharge will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gene F Kwan, MD MPH, Principal Investigator — Boston Medical Center, Cardiovascular Medicine
Locations (1):
- Zanmi Lasante/Hôpital Universitaire de Mirebalais, Mirebalais, Haiti

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT05091710/ICF_000.pdf